CLINICAL TRIAL: NCT02190825
Title: Safety and Efficacy Study of the NeuGuide Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pop Medical Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD0040
Record Dates: First submitted 2014-07-09; First posted 2014-07-15 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

INTERVENTIONS:
Device: NeuGuide device — The NeuGuideTM device is indicated for anchoring sutures to ligaments of the pelvic floor

SUMMARY:
This study aims to investigate the safety, efficacy, peri and postoperative complications, and patient satisfaction of sacro-spinous ligament fixation (SSLF) for the management of pelvic organ prolapse (POP).

Prolapse staging for all subjects in this study will be performed according to the POP-Q staging system.

Ultrasound examinations for all subjects in this study are subjected to the surgeon need and will be performed if required by qualified personnel

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-80 years old
* POP-Q stage III prolapse or higher
* Scheduled to undergo a POP Surgery and has agreed to undergo it using the NeuGuideTM device
* Patient is willing to return for follow-up evaluation and fill questionnaires as indicated on study protocol
* No exclusion criteria fulfilled

Exclusion Criteria:

* Diagnosis of reproductive tract anomalies
* Prior pelvic radiation therapy or any malignancy
* Inability to complete written questionnaires.
* Women with significant Pelvic Inflammatory Disease (PID) history
* Women with known allergy to Nickel or Nitinol

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Stage of pelvic floor prolapse as defined by POP-Q score | 6 months
Complications (SAE, AE) | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Wolfson Medical Center, Bat Yam
  - Hadassah Medical Center, Jerusalem